CLINICAL TRIAL: NCT04275687
Title: Thoracic Re-irradiation For Locoregionally Recurrent Non-small Cell Lung Cancer Using Hypofractionated Technique.
Brief Title: Thoracic Re-irradiation For Locoregionally Recurrent Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO1057
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Loco-regionally Recurrent NSCLC After Thoracic Radiotherapy
Keywords: loco-regionally recurrent non-small cell lung cancer; thoracic irradiation; hypofraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- thoracic irradiation (Experimental): For peripherally located recurrent tumors, stereotactic body radiation therapy is used at 5000-6000 cGy in 10 fractions.
  For centrally located recurrent tumors, adaptive hypofractionated radiation is used: Patients are irradiated at 3000-4000cGy in 6-10 daily fractions in the first course. After a four-week interval, patients who have non-progressive disease and an adequate pulmonary function undergo adaptive re-planning, and are irradiated at 2400-3500cGy in 4~7 daily fractions as a boost. Concurrent chemotherapy consists of weekly docetaxel and nedaplatin.
  Interventions: Radiation: thoracic irradiation; Drug: Concurrent chemotherapy

INTERVENTIONS:
Radiation: thoracic irradiation — For peripherally located recurrent tumors, stereotactic body radiation therapy is used at 5000-6000 cGy in 10 fractions.
  For centrally located recurrent tumors, adaptive hypofractionated radiation is used: Patients are irradiated at 3000-4000cGy in 6-10 daily fractions in the first course. After a four-week interval, patients who have non-progressive disease and an adequate pulmonary function undergo adaptive re-planning, and are irradiated at 2400-3500cGy in 4~7 daily fractions as a boost.
Drug: Concurrent chemotherapy — For centrally located recurrent tumors, concurrent chemotherapy consists of weekly docetaxel and nedaplatin.

SUMMARY:
This prospective phase II study is to assess the efficacy and safety of thoracic re-irradiation for locoregionally recurrent non-small cell lung cancer using hypofractionated technique.

DETAILED DESCRIPTION:
This prospective phase II study is to assess the efficacy and safety of thoracic re-irradiation for locoregionally recurrent non-small cell lung cancer using hypofractionated technique.

1. For peripherally located recurrent tumors, stereotactic body radiation therapy is used at 5000-6000 cGy in 10 fractions.
2. For centrally located recurrent tumors, adaptive hypofractionated radiation is used: Patients are irradiated at 3000-4000cGy in 6-10 daily fractions in the first course. After a four-week interval, patients who have non-progressive disease and an adequate pulmonary function undergo adaptive re-planning, and are irradiated at 2400-3500cGy in 4~7 daily fractions as a boost. Concurrent chemotherapy consists of weekly docetaxel and nedaplatin.

ELIGIBILITY:
Inclusion Criteria:

* loco-regionally recurrent NSCLC after thoracic radiotherapy (confirmed by pathology or continuous enhanced CT imaging);
* chemotherapy, targeted or immunotherapy are allowed before enrollment;
* >=6 months from previous chest radiotherapy;
* presence of measurable disease according to RECIST criteria;
* ECOG performance score is 0-1;
* organ and bone marrow functions meet the following criteria:

  * forced expiratory volume in 1 second (FEV1) ≥ 0.8L;
  * percentage-predicted single-breath carbon monoxide diffusing capacity (DLCO %) > 60%;
  * absolute neutrophil count ≥1.5×10^9/L;
  * platelet ≥80×10^9/L;
  * hemoglobin ≥9.0g/dL;
  * serum creatinine clearance was ≥50 mL/min calculated based on the Cockcroft-Gault formula
  * serum bilirubin ≤1.5 times normal upper limit (ULN)
  * AST and ALT≤2.5 times ULN

Exclusion Criteria:

* previous or concurrent with other malignant tumors, except for non-melanoma of the skin or carcinoma in situ of the cervix;
* loco-regional recurrence with distant metastasis;
* any other disease or condition contradicted to radiotherapy (e.g., active infection, within 6 months after myocardial infarction, symptomatic heart disease, including unstable angina, congestive heart failure or uncontrolled arrhythmia, immunosuppressive therapy);
* women who are pregnant or breastfeeding, women who have not undergone a pregnancy test (within 14 days before first administration), and women who are pregnant;
* pregnancy, lactation, or fertility but no contraceptive measures;
* those with bleeding tendency;
* participate in other clinical trials within 30 days before enrollment;
* drug and other drug addiction, chronic alcoholism and AIDS patients;
* having uncontrollable seizures or loss of self-control due to psychosis;
* a history of severe allergies;
* participants considered unfit to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2 years

SECONDARY OUTCOMES:
Local Control | 2 Years
Incidence of Grade ≥3 pulmonary toxicity/esophageal toxicity | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Prof., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Pfister DG, Johnson DH, Azzoli CG, Sause W, Smith TJ, Baker S Jr, Olak J, Stover D, Strawn JR, Turrisi AT, Somerfield MR; American Society of Clinical Oncology. American Society of Clinical Oncology treatment of unresectable non-small-cell lung cancer guideline: update 2003. J Clin Oncol. 2004 Jan 15;22(2):330-53. doi: 10.1200/JCO.2004.09.053. Epub 2003 Dec 22. No abstract available. PMID 14691125
- [Background] Goldstraw P, Chansky K, Crowley J, Rami-Porta R, Asamura H, Eberhardt WE, Nicholson AG, Groome P, Mitchell A, Bolejack V; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee, Advisory Boards, and Participating Institutions; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee Advisory Boards and Participating Institutions. The IASLC Lung Cancer Staging Project: Proposals for Revision of the TNM Stage Groupings in the Forthcoming (Eighth) Edition of the TNM Classification for Lung Cancer. J Thorac Oncol. 2016 Jan;11(1):39-51. doi: 10.1016/j.jtho.2015.09.009. PMID 26762738
- [Background] Curran WJ Jr, Paulus R, Langer CJ, Komaki R, Lee JS, Hauser S, Movsas B, Wasserman T, Rosenthal SA, Gore E, Machtay M, Sause W, Cox JD. Sequential vs. concurrent chemoradiation for stage III non-small cell lung cancer: randomized phase III trial RTOG 9410. J Natl Cancer Inst. 2011 Oct 5;103(19):1452-60. doi: 10.1093/jnci/djr325. Epub 2011 Sep 8. PMID 21903745
- [Background] Milton DT, Miller VA. Advances in cytotoxic chemotherapy for the treatment of metastatic or recurrent non-small cell lung cancer. Semin Oncol. 2005 Jun;32(3):299-314. doi: 10.1053/j.seminoncol.2005.02.011. PMID 15988685
- [Background] Noble J, Ellis PM, Mackay JA, Evans WK; Lung Cancer Disease Site Group of Cancer Care Ontario's Program in Evidence-based Care. Second-line or subsequent systemic therapy for recurrent or progressive non-small cell lung cancer: a systematic review and practice guideline. J Thorac Oncol. 2006 Nov;1(9):1042-58. PMID 17409993
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Kruser TJ, McCabe BP, Mehta MP, Khuntia D, Campbell TC, Geye HM, Cannon GM. Reirradiation for locoregionally recurrent lung cancer: outcomes in small cell and non-small cell lung carcinoma. Am J Clin Oncol. 2014 Feb;37(1):70-6. doi: 10.1097/COC.0b013e31826b9950. PMID 23357968
- [Background] Vyfhuis MAL, Rice S, Remick J, Mossahebi S, Badiyan S, Mohindra P, Simone CB 2nd. Reirradiation for locoregionally recurrent non-small cell lung cancer. J Thorac Dis. 2018 Aug;10(Suppl 21):S2522-S2536. doi: 10.21037/jtd.2017.12.50. PMID 30206496
- [Background] Kong FM, Ten Haken RK, Schipper MJ, Sullivan MA, Chen M, Lopez C, Kalemkerian GP, Hayman JA. High-dose radiation improved local tumor control and overall survival in patients with inoperable/unresectable non-small-cell lung cancer: long-term results of a radiation dose escalation study. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):324-33. doi: 10.1016/j.ijrobp.2005.02.010. PMID 16168827
- [Background] Schild SE, McGinnis WL, Graham D, Hillman S, Fitch TR, Northfelt D, Garces YI, Shahidi H, Tschetter LK, Schaefer PL, Adjei A, Jett J. Results of a Phase I trial of concurrent chemotherapy and escalating doses of radiation for unresectable non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):1106-11. doi: 10.1016/j.ijrobp.2006.02.046. Epub 2006 May 26. PMID 16730134
- [Background] Reyngold M, Wu AJ, McLane A, Zhang Z, Hsu M, Stein NF, Zhou Y, Ho AY, Rosenzweig KE, Yorke ED, Rimner A. Toxicity and outcomes of thoracic re-irradiation using stereotactic body radiation therapy (SBRT). Radiat Oncol. 2013 Apr 25;8:99. doi: 10.1186/1748-717X-8-99. PMID 23617949
- [Background] Spoelstra FO, Pantarotto JR, van Sornsen de Koste JR, Slotman BJ, Senan S. Role of adaptive radiotherapy during concomitant chemoradiotherapy for lung cancer: analysis of data from a prospective clinical trial. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1092-7. doi: 10.1016/j.ijrobp.2008.12.027. Epub 2009 Mar 26. PMID 19327915
- [Background] Gielda BT, Marsh JC, Zusag TW, Faber LP, Liptay M, Basu S, Warren WH, Fidler MJ, Batus M, Abrams RA, Bonomi P. Split-course chemoradiotherapy for locally advanced non-small cell lung cancer: a single-institution experience of 144 patients. J Thorac Oncol. 2011 Jun;6(6):1079-86. doi: 10.1097/JTO.0b013e3182199a7c. PMID 21532501
- [Background] Furuse K, Fukuoka M, Kawahara M, Nishikawa H, Takada Y, Kudoh S, Katagami N, Ariyoshi Y. Phase III study of concurrent versus sequential thoracic radiotherapy in combination with mitomycin, vindesine, and cisplatin in unresectable stage III non-small-cell lung cancer. J Clin Oncol. 1999 Sep;17(9):2692-9. doi: 10.1200/JCO.1999.17.9.2692. PMID 10561343
- [Background] Belani CP, Choy H, Bonomi P, Scott C, Travis P, Haluschak J, Curran WJ Jr. Combined chemoradiotherapy regimens of paclitaxel and carboplatin for locally advanced non-small-cell lung cancer: a randomized phase II locally advanced multi-modality protocol. J Clin Oncol. 2005 Sep 1;23(25):5883-91. doi: 10.1200/JCO.2005.55.405. Epub 2005 Aug 8. PMID 16087941
- [Background] Albain KS, Swann RS, Rusch VW, Turrisi AT 3rd, Shepherd FA, Smith C, Chen Y, Livingston RB, Feins RH, Gandara DR, Fry WA, Darling G, Johnson DH, Green MR, Miller RC, Ley J, Sause WT, Cox JD. Radiotherapy plus chemotherapy with or without surgical resection for stage III non-small-cell lung cancer: a phase III randomised controlled trial. Lancet. 2009 Aug 1;374(9687):379-86. doi: 10.1016/S0140-6736(09)60737-6. Epub 2009 Jul 24. PMID 19632716
- [Background] Vokes EE, Herndon JE 2nd, Kelley MJ, Cicchetti MG, Ramnath N, Neill H, Atkins JN, Watson DM, Akerley W, Green MR; Cancer and Leukemia Group B. Induction chemotherapy followed by chemoradiotherapy compared with chemoradiotherapy alone for regionally advanced unresectable stage III Non-small-cell lung cancer: Cancer and Leukemia Group B. J Clin Oncol. 2007 May 1;25(13):1698-704. doi: 10.1200/JCO.2006.07.3569. Epub 2007 Apr 2. PMID 17404369
- [Background] Saunders M, Dische S, Barrett A, Harvey A, Griffiths G, Palmar M. Continuous, hyperfractionated, accelerated radiotherapy (CHART) versus conventional radiotherapy in non-small cell lung cancer: mature data from the randomised multicentre trial. CHART Steering committee. Radiother Oncol. 1999 Aug;52(2):137-48. doi: 10.1016/s0167-8140(99)00087-0. PMID 10577699